CLINICAL TRIAL: NCT07146087
Title: Allogeneic Mesenchymal Stem Cell-Derived Exosome Therapy for Progressive Multiple Sclerosis
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow enrolment of participants
Sponsor: Biocells Medical (Industry)
Responsible Party: Principal Investigator, Andrei Peskau, Specialist in regenerative medicine, Biocells Medical
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: Bio120002
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: sclerosis; multiple sclerosis; MSC
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSC-Derived Exosomes (Experimental): Participants receive intravenous infusions of allogeneic mesenchymal stem cell (MSC)-derived exosomes every 12 weeks for 48 weeks (total of 4 infusions) in addition to their stable background MS therapy (if any).
  Interventions: Biological: MSC-Derived Exosomes
- Normal Saline (Placebo Comparator): Participants receive intravenous infusions of 0.9% sodium chloride (saline) matched in volume, appearance, and schedule to the experimental arm, in addition to their stable background MS therapy (if any).
  Interventions: Biological: Placebo (Normal Saline)

INTERVENTIONS:
Biological: MSC-Derived Exosomes — Purified, sterile, acellular extracellular vesicles (exosomes) isolated from culture supernatant of GLP-manufactured allogeneic human bone-marrow-derived MSCs. Release criteria include particle size distribution 30-150 nm (nanoparticle tracking analysis), particle count, sterility/endotoxin testing, mycoplasma negative, and predefined protein/marker profile (e.g., CD9/CD63/CD81 positive).
  Arms: MSC-Derived Exosomes
Biological: Placebo (Normal Saline) — 0.9% sodium chloride solution matched to the experimental product in volume, appearance, infusion set-up, and administration procedures.
  Arms: Normal Saline

SUMMARY:
The goal of this clinical trial is to learn if intravenous infusion of allogeneic mesenchymal stem cell (MSC)-derived exosomes can slow disability progression and improve neurological function in adults with progressive multiple sclerosis (MS). The trial will also evaluate the safety and tolerability of repeated exosome infusions.

The main questions it aims to answer are:

Does MSC-derived exosome therapy reduce disability progression as measured by the Expanded Disability Status Scale (EDSS)?

Does MSC-derived exosome therapy decrease neuroinflammation and brain lesion burden compared with placebo?

Researchers will compare participants who receive MSC-derived exosome therapy to those who receive placebo (saline infusion) to see if the treatment improves clinical and biological outcomes.

Participants will:

Receive either MSC-derived exosome infusions or placebo infusions every 3 months for 1 year (4 total infusions)

Undergo clinical assessments (neurological exams, EDSS scoring, neurocognitive testing)

Provide blood and cerebrospinal fluid samples for biomarker analysis

Have MRI scans to evaluate lesion load and brain volume

Complete questionnaires on quality of life and daily functioning

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Diagnosis of progressive multiple sclerosis (primary or secondary) confirmed
3. EDSS score 3.0-6.5.

Exclusion Criteria:

1. Relapse or corticosteroid treatment within 3 months before screening.
2. Other significant neurological or autoimmune disorders.
3. Active infection, malignancy, or uncontrolled systemic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score | 24 months from the day of administration
  Unit of measure: points (range: 0-10; higher scores indicate worse disability).

SECONDARY OUTCOMES:
Change in T2 lesion load and brain atrophy | 24 months after the first administration
  On MRI Unit: number and volume of lesions (mm³).
Change in neurocognitive performance | 24 months after first administration
  Assessed via Symbol Digit Modalities Test (SDMT). Unit: score (range: 0-110; higher scores mean better cognition).

CONTACTS AND LOCATIONS:
Locations (1):
- Biocells Medical, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No